CLINICAL TRIAL: NCT06557330
Title: HM-225: Measurable Residual Disease (MRD) Guided De-intensification of Bendamustine/Rituximab (BR) for Indolent Non-Hodgkin Lymphoma
Brief Title: MRD Guided De-intensification of Bendamustine/Rituximab for Indolent Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Adaptive Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-1014, HM-225
Record Dates: First submitted 2024-08-09; First posted 2024-08-16 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma; Indolent Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bendamustine Hydrochloride; Rituximab; Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): This is a phase II pilot, single arm, open label study designed to assess the efficacy, safety, and feasibility of Measurable Residual Disease (MRD) adapted duration of BR for untreated or R/R iNHL (indolent non-hodgkin lymphoma). All patients will receive Bendamustine 90 mg/m2 IV on Days 1-2 and Rituximab 375 mg/m2 IV(BR) on Day 1 of each cycle. Each cycle will last 28 days. On day 1 of each cycle, patients will receive Rituximab before Bendamustine, and CBC (complete blood count), CMP (comprehensive metabolic panel) will be obtained to capture any hematologic toxicities as well as clonoSEQ testing to determine MRD status. After completing Cycle 3, imaging results (with confirmatory biopsy if applicable) and the clonoSEQ MRD testing results obtained from ctDNA (blood collection) will determine whether patients will receive Cycles 5 and 6 of Bendamustine and Rituximab (BR).
  Interventions: Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine will be administered as 10 minute IV infusion at 90 mg/m2 (drug dose calculation is based on treatment day weight) on days 1 and 2 for 4-6 cycles (number of cycles determined per treatment design). Subjects will be dosed every 28 days. Ondansetron 16 mg IV is given as premedication per institutional guidelines. Dose modifications will be determined based on renal and hepatic function. Subjects should be carefully monitored for infusion reactions during Bendamustine administration. If an acute infusion reaction is noted, subjects should be managed according to institutional guidelines. Doses of Bendamustine may be interrupted, delayed, or discontinued depending on how well the subject tolerates the treatment based on physician discretion.
  Other Names: cytostasan; belrapzo; treanda; vivimusta
Drug: Rituximab — Rituximab will be administered as an IV infusion at 375 mg/m2 (longer for the first dose) (drug dose calculation is based of treatment day weight) on day 1 for 4-6 cycles (number of cycles determined per treatment design). Infusion rate will be determined as per institutional standards. Subjects will be dosed every 28 days. Diphenhydramine 50 mg IV and acetaminophen 650 mg are required to be given to the subjects within 30 minutes prior to Rituximab dose. There are no dose modifications recommended with Rituximab. If an acute infusion reaction is noted, subjects should be managed according to institutional guidelines. Doses of Rituximab may be interrupted, delayed, or discontinued depending on how well the subject tolerates the treatment.
  Other Names: riabni; Rituxan; Ruxience; Truxima; Azulfidine

SUMMARY:
This is a phase II pilot, single arm, open label study designed to assess the efficacy, safety, and feasibility of MRD adapted duration of BR for untreated or R/R iNHL.

DETAILED DESCRIPTION:
This is a phase II pilot, single arm, open label study designed to assess the efficacy, safety, and feasibility of MRD adapted duration of BR for untreated or R/R iNHL.

All patients with untreated or R/R (not previously treated with Bendamustine) iNHL (Follicular Lymphoma (Grade 1-3a2), Marginal Zone Lymphoma, Lymphoplasmacytic Lymphoma) are candidates for this trial. Patients requiring treatment per treating physician's discretion are eligible for the trial.

Patients who recently started on and received two cycles of Bendamustine at 90 mg/m2 dose with Ritxumab 375 mg/m2 are also eligible for this trial. For these patients, C2D1 BR should be no more than 14 days prior to the time of study enrollment (i.e. enrollment no later than C2D14). Patients who have received two cycles of 90mg/m2 Bendamustine dose with Rituximab 375 mg/m2 can enter the study and initiate cycle 3 once pre-screening and screening procedures have been completed.

ELIGIBILITY:
Inclusion Criteria:

Patients must have pathologically confirmed:

* indolent Non-Hodgkin Lymphoma, consistent with one of the below diagnoses:
* Follicular Lymphoma (Grade 1-3a)
* Marginal Zone Lymphoma
* Lymphoplasmacytic Lymphoma

Patient may be treatment naïve or relapsed/refractory without having received prior Bendamustine or patients recently started on Bendamustine 90 mg/m2 with Rituximab 375 mg/m2 are eligible if C2D1 BR is no more than 14 days prior to enrollment and they otherwise meet eligibility criteria

* Age > 18 years
* ECOG performance status 0-2

Patients must have normal organ and marrow function as defined below:

* Absolute Neutrophil Count >1000mm3 and Hemoglobin >8 g/dL (unless due to bone marrow involvement by lymphoma)
* Total bilirubin > 1.5x upper limit of normal (patients with Gilbert's syndrome can have total bilirubin up to 3x upper normal limit)
* Aspartate aminotransferase/ alanine aminotransferase (serum glutamic-oxaloacetic transaminase/ serum glutamic-pyruvic transaminase) < 5 times institutional normal limits
* Creatinine clearance > 30 Ml/min

Exclusion Criteria:

* Radiation or systemic treatment for lymphoma within the past 28 days prior to cycle 1 day 1 of BR.
* Patients with pathologically confirmed transformed lymphoma, including diffuse large B cell lymphoma or other high grade lymphomas
* Patients on active treatment for second malignancy with the exception of endocrine therapy for non-metastatic breast cancer, hormone therapy for prostate cancer, or local treatment for non-melanoma skin cancer.
* Pregnant or breast-feeding. Refer to section 5.4 for further detail.
* Failure to identify a dominant clonal sequence with ClonoSEQ from pre-treatment specimen or inadequate tissue for testing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-09-29 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
PFS Evaluation | 2 years
  To evaluate the 2-year progression free survival (PFS) for patients treated with Bendamustine and Rituximab (BR) with measurable residual disease directed (MRD) duration of therapy.
Statistical PFS | 2 years
  The proportion (p) of patients who are progression-free and are alive at 2 years from the initiation of treatment using Lugano Criteria.

SECONDARY OUTCOMES:
Secondary Outcome Measure | 2 years
  Assess additional clinical outcomes including overall survival (OS),
Measurable Residual Disease Evaluation | 2 years
  To determine the rate of MRD (minimal residual disease) negativity at end of treatment and at 2 years post-treatment
Adverse Event assessment | 2 years
  Assess adverse effects of treatment
Overall Survival Assessment | 2 years
  OS, defined as time from initiation of study treatment until death, or the end of follow-up, whichever occurs first. Patients who are still alive at the end of follow-up will be considered censored.
Measurable Residual Disease Negativity | 2 years
  To evaluate MRD negativity rate at the end of treatment and at 2 years post-treatment.
Rate of 3+ adverse events | 2 years
  The rate of grade 3+ adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.The rate of grade 3+ adverse events as assessed by CTCAE v5.0.

OTHER OUTCOMES:
Exploratory Outcome Measures | 2 years
  Assess and compare measurable residual disease (MRD) sensitivity of both circulating tumor DNA (ctDNA) and circulating tumor cells (CTC), both being obtained at baseline, after each cycle, and during follow up
Measurable Residual Disease (MRD) | 2 years
  Assess MRD level, both ctDNA and circulating tumor cell (CTC) testing, after each cycle of Bendamustine and Rituximab (BR) and correlate with Progression Free Survival (PFS)
Progression Free Survival (PFS) for Measurable Residual Disease (MRD) | 2 years
  To evaluate PFS for patients with low level detectable MRD (10^-4 to 10^-6) after 3 cycles of Bendamustine and Rituximab
Measurable Residual Disease (MRD) to guide indolent lymphoma treatment evaluation | 2 years
  Evaluate feasibility of using MRD to guide treatment for indolent lymphoma
Measurable Residual Disease (MRD) failure rate | 2 years
  Determine MRD test baseline failure rate from ctDNA and Circulating Tumor Cell (CTC) testing
Infection occruance | 2 years
  Assess occurrence of infection of any grade
Secondary malignancy occurrence | 2 years
  Assess occurrence of secondary malignancy
Ntural Killer and T cell reconstitution | 2 years
  Assess the rate of NK (natural kiler) cell and T cell subset reconstitution after Bendamustine and Rituximab; distinguish if there is difference between shorter/longer treatment regimens
Quality Life Assessment | 2 years
  Assess differences in quality of life based on Functional Assessment of Cancer Therapy (FACT-Lym) questionnaire between patients who received varying lengths of treatment.
Baseline Proliferative Rate | 2 years
  Correlation of baseline proliferative rate

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Messmer, Principal Investigator — Fox Chase Cancer Center